CLINICAL TRIAL: NCT01515150
Title: Management of Patients With Uncomplicated Diverticulitis as Out-patient and Without Antibiotics
Brief Title: The Out-patient, Non Antibiotic Management of Patients With Acute Uncomplicated Colonic Diverticulitis
Acronym: P-VOD
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: P-VOD
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Colonic Diverticulitis
Keywords: diverticulitis; Out-patient management; Antibiotics
MeSH Terms: conditions — Diverticulitis, Colonic; Diverticulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Out-patients in diverticulitis: All patient with acute uncomplicated diverticulitis how accept participation in the study will be enrolled in the study.

SUMMARY:
Previous multicentre study NCT 01008488 indicates that a patient with CT-proven uncomplicated diverticulitis has a very low risk (1.4%) of developing severe complications such as perforations or abscesses. The question is whether or not hospitalization is necessary, and if patients in that case could return home without antibiotics.

The purpose of this study is to evaluate if out-patients managements in uncomplicated colonic diverticulitis is possible without readmission or complications.

DETAILED DESCRIPTION:
At the emergency room all patients with computed tomography verified acute uncomplicated diverticulitis will be asked about participation in the study. If They accept the participation, They will be send home with pain relief medicine. Every morning a nurse from our colorectal unit call the patient asking about the condition. The patients will have a visit at the surgery unit within 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age above 18 years, acute abdominal pain (Duration< 3 days), abdominal tenderness, elevated inflammatory parameters, CT- scan sign of uncomplicated diverticulitis(without sign of abscess or free air).

Exclusion Criteria:

* diffuse peritonitis sepsis or abscess, drying Patients who are unable to intake of fluids orally, severe pain with need of repeated parenteral morphine treatment, immunological deficient patients incl. steroid treatment, pregnancy, dementia, patients who need hospitalization of other reasons

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CT- scan varified acute uncomplicated diverticulitis how are abel to underwent out-patients managment
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of admission and complications among participant within three months follow-up. | Three months

SECONDARY OUTCOMES:
To evaluate reason of hospital admission, late complications, need of bowel rest and costs | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Mats Enlund, Ass. Prof, Study Chair — Centre of Clinical Research of Uppsala University, Västmanlands Hospital Västerås
Locations (1):
- Colorectal unit, department of surgery Västmanland Hospital Västerås, Västerås, Västmanland County, Sweden